CLINICAL TRIAL: NCT06506097
Title: Community-viable Family-school Partnership Intervention for Children With Social-communication Deficits in Early Childhood Education
Brief Title: Family-school Partnership Intervention for Early Childhood Education
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas, Denton, TX (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Michael Siller, Associate Professor, University of North Texas, Denton, TX
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7R21HD105168-02 (NIH)
Record Dates: First submitted 2024-06-14; First posted 2024-07-17 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; preschool; Naturalistic Developmental Behavioral Intervention; education; parent
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Uncontrolled (pre-post) clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Family-school Partnership Intervention (FSPI) (Experimental): Participants include 20 non-teaching support staff (1-2 per program), 30 lead teachers (2-4 per program), and 60 children with social-communication deficits (two per teacher). FSPI creates new opportunities for teachers to partner with families, particularly parents of children with social-communication vulnerabilities. Specifically, teachers will be provided with a curriculum, training, and resources to engage two families from their classroom in three FSPI Playgroup meetings, scheduled over the course of the current school year. During each playgroup, teaches will help parents practice simple strategies for promoting communication during familiar routines such as play, book reading, preparing a snack, or completing a simple chore.
  Interventions: Behavioral: Family-school Partnership Intervention (FSPI)

INTERVENTIONS:
Behavioral: Family-school Partnership Intervention (FSPI) — FSPI includes implementation activities across multiple levels.
  FSPI Planning Team Meetings will be held monthly to plan project activities, practice staff and parent coaching strategies, and troubleshoot implementation challenges.
  FSPI Staff Training (3 hours) will be provided during a single professional development day (3 hours), and attended by members of the FSPI Planning Team and teachers.
  FSPI Playgroups. Over the course of the school year, each parent-child dyad will be invited to participate in three FSPI Playgroup events. Typically, teachers from two classrooms will collaborate in hosting playgroup events, and each playgroup will be attended by four parent-child dyads (i.e., two per classroom). Teachers will be provided with a curriculum and learning outcomes to target.
  FSPI Debrief Meetings are held after each FSPI Playgroup to debrief, reflect, and improve FSPI implementation.

SUMMARY:
Strategies for creating and maintaining reciprocal partnerships between teachers and parents are considered essential elements of developmentally appropriate practice in early childhood education (ECE). Particularly for children who are high-risk for behavioral, developmental, or mental health problems, effective partnerships between family and preschool are essential for promoting optimal classroom participation and learning outcomes. The current study is an uncontrolled (pre-post) feasibility trial of Family-School Partnership Intervention (FPSI). FSPI was developed using stakeholder input, is delivered by existing preschool staff, and aims to promote development and reduce barriers to learning among children with pre-clinical social-communication delays. FSPI integrates evidence-based practices (EBPs) from education (7 EBPs; National Association for the Education of Young Children) with clinical interventions for toddlers with autism spectrum disorder (ASD) (12 EBPs at the educator-parent level and 8 EBPs at the parent-child level; Naturalistic Developmental Behavioral Interventions). Data will be collected across 10 ECE programs. At each participating ECE program, research procedures will be completed during a single school year. Selected ECE programs will include public school, Head Start, and private preschool programs. Participants include 20 non-teaching support staff (1-2 per program; e.g., director, principal, education-coordinator), 30 lead teachers (2-4 per program), and 60 children with social-communication deficits (two per teacher). Data collection will focus on feasibility data (enrollment, attendance, attrition, data completion), observational measures of implementation fidelity (at the educator-parent and parent-child level), and mixed methods to evaluate educator and parent acceptability and satisfaction and identify implementation drivers/barriers. This research will prepare a large, multi-site hybrid trial to evaluate the effectiveness of FSPI for promoting social-communication skills and kindergarten readiness, in addition to factors that mediate the relation between FSPI delivery and fidelity (implementation drivers/barriers).

ELIGIBILITY:
Inclusion Criteria:

* currently attending classroom of participating preschool teacher.
* nominated by teacher as child with elevated levels of social-communication challenges

Exclusion Criteria:

* n/a

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility benchmark - Enrollment | Through study completion, an average of 1 year
  Throughout we will collect administrative data on enrollment. Data will be judged against pre-specified feasibility criteria: Enrollment (20 non-teaching staff, 30 teachers, 60 parents) will meet 100% of target.
Feasibility benchmark - FSPI Completion | Through study completion, an average of 1 year
  Throughout we will collect administrative data on attrition. Data will be judged against pre-specified feasibility criteria: % of parents completing the intervention. Benchmarks: >80% for FSPI completion, >75% for session attendance (parents), and >80% for measure completion (staff, parents).
Feasibility benchmark - Session Attendance | Through study completion, an average of 1 year
  Throughout we will collect administrative data on session attendance. Data will be judged against pre-specified feasibility criteria: % of sessions completed by preschool staff and parents. Benchmarks: >75% for session attendance.
Feasibility benchmark - Measure Completion | Through study completion, an average of 1 year
  Throughout we will collect administrative data on data collection components. Data will be judged against pre-specified feasibility criteria: % of measures completed by preschool staff and parents: Benchmarks: >80%.

CONTACTS AND LOCATIONS:
Locations (1):
- UNT, Denton, Texas, United States

IPD SHARING:
Plan to Share IPD: No